CLINICAL TRIAL: NCT05665998
Title: Brain Controlled Spinal Cord Stimulation in Participants With Cervical Spinal Cord Injury for Upper Limb Rehabilitation (UP2)
Brief Title: Brain Controlled Spinal Cord Stimulation in Participants With Cervical Spinal Cord Injury for Upper Limb Rehabilitation
Acronym: UP2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Principal Investigator, Jocelyne Bloch, Certified neurosurgeon, head of functional neurosurgery, Ecole Polytechnique Fédérale de Lausanne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UP2
Record Dates: First submitted 2022-12-14; First posted 2022-12-27 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Cervical Spinal Cord Injury; Tetraplegia
Keywords: Spinal cord stimulation; Brain computer interface; Brain spine interface
MeSH Terms: conditions — Quadriplegia

STUDY DESIGN:
Intervention Model Description: single-site, single-arm, non-blinded, non-randomized, interventional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARC-BSI Cervical Rehabilitation (Experimental): Implantation of a neuroprosthetics system composed of an electrocorticography acquisition system (WIMAGINE) and a cervical epidural electrical spinal cord stimulation system (ARC-IM) to restore voluntary arm movements in participants with SCI.
  Interventions: Device: ARC-BSI Cervical system

INTERVENTIONS:
Device: ARC-BSI Cervical system — Unilateral implantation of a 64 channel - ECoG array over the sensory motor cortex combined with an implantation of 32 channel spinal cord stimulation system over the cervical region. The system decodes the motor attempts of the participant and translates those intentions into modulation of electrical stimulation.

SUMMARY:
Cervical spinal cord stimulation can elicit arm and hand movements through recruitment of proprioceptive neurons in the dorsal roots. In participants with cervical spinal cord injury, the spare roots bellow the lesion can be used to reactivate motor function. Decoding of motor intentions can be achieved through implantable electrocorticography (ECoG) devices.

In this study, the investigators will use an investigational system using ECoG signal recording over the motor cortex to drive muscle specific electrical epidural spinal cord stimulation (EES). The investigators will assess the safety and preliminary efficacy of this system in 3 participants.

DETAILED DESCRIPTION:
In a current first-in-human clinical trial, called STIMO, Electrical Epidural Spinal Stimulation (EES) is applied to enable individuals with chronic severe spinal cord injury (SCI) to complete intensive locomotor neurorehabilitation training. In this clinical feasibility study, EES triggered an immediate enhancement of walking function, and was integrated in an intensive neurorehabilitation program. This therapy improved leg motor control and triggered neurological recovery in individuals with severe SCI to a certain extent (Wagner et al. 2018, Kathe et al. 2022).

Concurrently, preclinical and clinical evidence demonstrated a similar recruitment of upper limb muscles through cervical spinal cord stimulation, re-triggering arm movements after paralysis. The spatial and temporal modulation of the electrical stimulation can selectively activate muscle groups towards a specific function.

Clinatec (CEA, Grenoble, France) has developed an implantable electrocorticogram (ECoG) recording device with a 64-channel epidural electrode array capable of recording electrical signals from the motor cortex for an extended period and with a high signal to noise ratio. This ECoG-based system allowed tetraplegic patients to control an exoskeleton (Clinicaltrials.gov, NCT 02550522) with up to 8 degrees of freedom for the upper limb control (Benabid et al., 2019). This device has been implanted in 4 individuals so far; one of them has been using this system both at the hospital and at home for more than 3 years.

Another ongoing clinical study: STIMO-BSI (Brain Spine Interface) (Clinicaltrials.gov: NTC04632290), is combining the EES and ECoG technology to allow leg motor control in patients with chronic SCI through the decoding of cortical signals.

In this study, the investigators will test the safety and preliminary efficacy of ECoG-controlled EES in individuals with cervical SCI and establish a direct bridge between the participants' motor intention and the spinal cord below the lesion, which could restore voluntary control of arm movements as well as promote neurological recovery when combined with neurorehabilitation.

ELIGIBILITY:
* Must provide Informed Consent as documented by signature (Appendix Informed Consent Form),
* Must be at least 18 years old and no older than 75 years old at the time of enrolment,
* Must be suffering from non-progressive traumatic cervical spinal cord injury,
* Must be graded A, B, C, or D in the American Spinal Injury Association (ASIA) Impairment Scale (AIS) classification,
* Must have completed primary standard of care rehabilitation,
* Must be severely impaired in his upper limb function as determined by the investigator,
* Must have sustained the injury at least 6 months before signing the consent form,
* Must be able to understand and interact with the study team in French or English,
* Must agree to comply in good faith with all conditions of the study and to attend all scheduled appointments,
* Must use safe contraception for women of childbearing capacity,
* Must not be pregnant nor breast feeding,
* Must not have history of severe autonomic dysreflexia,
* Must not have brain damage,
* Must not have history of epilepsy,
* Must not have spinal stenosis,
* Must not have gastrointestinal ulcers in the last five years,
* Must not have any psychological disorder,
* Must not have the intention to become pregnant during the course of the study,
* Must not be known or suspected of drug or alcohol abuse,
* Must not have participated in another clinical study using drugs or medical devices within the 30 days preceding and during the present study,
* Must not have previously been injected with stem cells in the spinal cord,
* Must not be the investigator himself, his/her family members, employees or other dependent persons,
* Must not have any unstable or significant medical condition that is likely to interfere with study procedures or likely to confound study endpoint evaluations as determined by the Investigator,
* Must not have any hematological disorders with increased risk for surgical intervention,
* Must not require ventilator support,
* Must not suffer from spinal cord injury from other etiology than traumatic (ischemic, tumoral, autoimmune, etc),
* Must not be subject to spasms that limit the ability of the subject to participate in the study training as determined by the investigator,
* Must not display spinal stenosis or post traumatic damage at location of implantation,
* Must not require the use of an intrathecal baclofen pump,
* Must not be implanted with a device such as pacemakers or defibrillators,
* Must not have any indication that would require an MRI,
* Must not suffer from congenital nor acquired upper limb abnormalities (affection of joints or bones).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Number of treatment-related serious adverse events (SAEs). | Through completion of the study 12 months

SECONDARY OUTCOMES:
Graded and Redefined Assessment of Strength Sensibility, and Prehension (GRASSP) score | 7 months
  0-232 points, higher score indicating better performance
Action Research Arm Test (ARAT) score | 7 months
  0-57 points, higher score indicating better performance
Capabilities of the Upper Extremity Test (CUE-T) | 7 months
  0-68 points, higher score indicating better performance
Range of Motion (in rad) | 7 months
Grasp force (in N) | 7 months
Pinch force (in N) | 7 months
International Standards for Neurological Classification of SCI (ISNCSCI) score | 7 months
  0-324 points, higher score indicating better function
Maximum voluntary contraction (in N.m) | 7 months
Somato-sensory evoked potential amplitude (in mV) | 7 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wagner FB, Mignardot JB, Le Goff-Mignardot CG, Demesmaeker R, Komi S, Capogrosso M, Rowald A, Seanez I, Caban M, Pirondini E, Vat M, McCracken LA, Heimgartner R, Fodor I, Watrin A, Seguin P, Paoles E, Van Den Keybus K, Eberle G, Schurch B, Pralong E, Becce F, Prior J, Buse N, Buschman R, Neufeld E, Kuster N, Carda S, von Zitzewitz J, Delattre V, Denison T, Lambert H, Minassian K, Bloch J, Courtine G. Targeted neurotechnology restores walking in humans with spinal cord injury. Nature. 2018 Nov;563(7729):65-71. doi: 10.1038/s41586-018-0649-2. Epub 2018 Oct 31. PMID 30382197
- [Background] Kathe C, Skinnider MA, Hutson TH, Regazzi N, Gautier M, Demesmaeker R, Komi S, Ceto S, James ND, Cho N, Baud L, Galan K, Matson KJE, Rowald A, Kim K, Wang R, Minassian K, Prior JO, Asboth L, Barraud Q, Lacour SP, Levine AJ, Wagner F, Bloch J, Squair JW, Courtine G. The neurons that restore walking after paralysis. Nature. 2022 Nov;611(7936):540-547. doi: 10.1038/s41586-022-05385-7. Epub 2022 Nov 9. PMID 36352232
- [Background] Rowald A, Komi S, Demesmaeker R, Baaklini E, Hernandez-Charpak SD, Paoles E, Montanaro H, Cassara A, Becce F, Lloyd B, Newton T, Ravier J, Kinany N, D'Ercole M, Paley A, Hankov N, Varescon C, McCracken L, Vat M, Caban M, Watrin A, Jacquet C, Bole-Feysot L, Harte C, Lorach H, Galvez A, Tschopp M, Herrmann N, Wacker M, Geernaert L, Fodor I, Radevich V, Van Den Keybus K, Eberle G, Pralong E, Roulet M, Ledoux JB, Fornari E, Mandija S, Mattera L, Martuzzi R, Nazarian B, Benkler S, Callegari S, Greiner N, Fuhrer B, Froeling M, Buse N, Denison T, Buschman R, Wende C, Ganty D, Bakker J, Delattre V, Lambert H, Minassian K, van den Berg CAT, Kavounoudias A, Micera S, Van De Ville D, Barraud Q, Kurt E, Kuster N, Neufeld E, Capogrosso M, Asboth L, Wagner FB, Bloch J, Courtine G. Activity-dependent spinal cord neuromodulation rapidly restores trunk and leg motor functions after complete paralysis. Nat Med. 2022 Feb;28(2):260-271. doi: 10.1038/s41591-021-01663-5. Epub 2022 Feb 7. PMID 35132264
- [Background] Larzabal C, Bonnet S, Costecalde T, Auboiroux V, Charvet G, Chabardes S, Aksenova T, Sauter-Starace F. Long-term stability of the chronic epidural wireless recorder WIMAGINE in tetraplegic patients. J Neural Eng. 2021 Sep 9;18(5). doi: 10.1088/1741-2552/ac2003. PMID 34425566
- [Background] Benabid AL, Costecalde T, Eliseyev A, Charvet G, Verney A, Karakas S, Foerster M, Lambert A, Moriniere B, Abroug N, Schaeffer MC, Moly A, Sauter-Starace F, Ratel D, Moro C, Torres-Martinez N, Langar L, Oddoux M, Polosan M, Pezzani S, Auboiroux V, Aksenova T, Mestais C, Chabardes S. An exoskeleton controlled by an epidural wireless brain-machine interface in a tetraplegic patient: a proof-of-concept demonstration. Lancet Neurol. 2019 Dec;18(12):1112-1122. doi: 10.1016/S1474-4422(19)30321-7. Epub 2019 Oct 3. PMID 31587955
- [Background] Lorach H, Charvet G, Bloch J, Courtine G. Brain-spine interfaces to reverse paralysis. Natl Sci Rev. 2022 Jan 18;9(10):nwac009. doi: 10.1093/nsr/nwac009. eCollection 2022 Oct. No abstract available. PMID 36196116